CLINICAL TRIAL: NCT04406441
Title: Patient-Clinic-Community Integration to Prevent Obesity Among Rural Preschool Children
Acronym: ENCIRCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Penn State University (Other); Iowa State University (Other); University of Nebraska (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0207
Record Dates: First submitted 2020-05-21; First posted 2020-05-28 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Obesity; Preventive Medicine; Mentoring; Food Supply
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Participants will attend regularly scheduled well child visits (WCV) that follow standard clinical guidelines. Well child visits will include review of history, age-appropriate measurements (height/length, weight, body mass index (BMI), blood pressure), sensory and developmental screenings, physical exam, immunizations, oral health review, and anticipatory guidance (preventive counseling).
- Patient Reported Outcome (Active Comparator): Arm 2 builds on the standard of care WCV by adding a patient reported outcome measure, the Family Nutrition and Physical Activity risk assessment, to inform family-centered preventative counseling during clinical care.
  Interventions: Behavioral: Patient Reported Outcome Well Child Visit
- Patient Reported Outcome + Food Care (Active Comparator): Participants will receive all Arm 2 components, in addition to be referred to both the Geisinger Wellness Program for a Parent Training Program and a grocery store nutritionist for a tour aligned with the Cooking Matters program.
  Interventions: Behavioral: Patient Reported Outcome Well Child Visit + Food Care

INTERVENTIONS:
Behavioral: Patient Reported Outcome Well Child Visit — Parents will complete the Family Nutrition and Physical Activity risk assessment (Patient Reported Outcome) prior to scheduled well child visit. Parent reported data is integrated into the child's electronic health record to inform the child's primary care provider and the provision of preventive counseling. The primary care provider documents preventive care provided.
  Arms: Patient Reported Outcome
Behavioral: Patient Reported Outcome Well Child Visit + Food Care — Adapted Parent Training Program will be delivered via telehealth (video or telephone) to parents by trained Wellness Coaches as 6 individual sessions, distributed throughout a 26-week intervention period. Cooking Matters grocery store tours will be delivered (in-person or virtual) to parents by trained grocery store nutritionists during the 26-week intervention period.
  Arms: Patient Reported Outcome + Food Care

SUMMARY:
The goal of this research study is to compare two enhancements to well-child visits at Geisinger designed to promote family-centered counseling for the prevention of obesity in a high-risk population of rural, lower income, preschool-aged children. Compared to the standard well-child visit, enhancements will offer advantages to obesity prevention, parent involvement in counseling, lifestyle behaviors, and food resource management.

ELIGIBILITY:
Inclusion Criteria:

* Age (20-months to 59-months, 29-days old)
* BMI-for-age and -sex >50th percentile based on WHO growth standards
* Parent commitment to participate in 18-month study
* Plans to attend scheduled WCV and recommended follow-up WCV in 12 months
* No plans to move or change health systems in 2 years
* Parent age > 18 years
* Parent is English-speaking
* Household is considered lower-income (i.e., eligible for or receiving Special Supplemental Nutrition Program for Women, Infants and Children [WIC], Supplemental Nutrition Assistance Program [SNAP], Temporary Assistance for Needy Families [TANF], Medicaid, or Children's Health Insurance Program [CHIP]) or screens positive for food insecurity.

Exclusion Criteria:

* Another child in family is participating
* Pre-existing medical exclusions (cancer, type 1 diabetes, major developmental delays such as autism)
* Parents with self-reported major depression will be excluded.

Ages: 20 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2040 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bailey-Davis, DEd, RD, Principal Investigator — Geisinger Clinic
Locations (1):
- Shawnee L Lutcher, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slusser W, Frankel F, Robison K, Fischer H, Cumberland WG, Neumann C. Pediatric overweight prevention through a parent training program for 2-4 year old Latino children. Child Obes. 2012 Feb;8(1):52-9. doi: 10.1089/chi.2011.0060. PMID 22799481
- [Background] Bailey-Davis L, Kling SMR, Wood GC, Cochran WJ, Mowery JW, Savage JS, Stametz RA, Welk GJ. Feasibility of enhancing well-child visits with family nutrition and physical activity risk assessment on body mass index. Obes Sci Pract. 2019 Apr 24;5(3):220-230. doi: 10.1002/osp4.339. eCollection 2019 Jun. PMID 31275595
- [Background] Bailey-Davis L, Moore AM, Poulsen MN, Dzewaltowski DA, Cummings S, DeCriscio LR, Hosterman JF, Huston D, Kirchner HL, Lutcher S, McCabe C, Welk GJ, Savage JS. Comparing enhancements to well-child visits in the prevention of obesity: ENCIRCLE cluster-randomized controlled trial. BMC Public Health. 2022 Dec 26;22(1):2429. doi: 10.1186/s12889-022-14827-w. PMID 36572870
- [Background] Potts BA, Wood GC, Bailey-Davis L. Agreement between parent-report and EMR height, weight, and BMI among rural children. Front Nutr. 2024 Mar 1;11:1279931. doi: 10.3389/fnut.2024.1279931. eCollection 2024. PMID 38496791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary Care Providers were the unit of randomization in this study. Parent/child dyads were enrolled and were assigned to one of the three study arms based on which provider they saw for their regular well-child visits. There were 105 providers trained and randomized, 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads. Below enrollment data reflects the randomization of the parent/child dyads.
Units Other Than Participants: Providers
Period: Overall Study
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Started | 1422; 34 Providers (Participants include 711 unique parents and 711 unique children that combined to form a total of 711 dyads.) | 1504; 35 Providers (Participants include 752 unique parents and 752 unique children that combined to form a total of 752 dyads.) | 1154; 36 Providers (Participants include 577 unique parents and 577 unique children that combined to form a total of 577 dyads.)
Parents | 711; 34 Providers | 752; 35 Providers | 577; 36 Providers
Children | 711; 34 Providers | 752; 35 Providers | 577; 36 Providers
Completed | 1422; 34 Providers (Participants include 711 unique parents and 711 unique children that combined to form a total of 711 dyads.) | 1504; 35 Providers (Participants include 752 unique parents and 752 unique children that combined to form a total of 752 dyads.) | 1154; 36 Providers (Participants include 577 unique parents and 577 unique children that combined to form a total of 577 dyads.)
Not Completed | 0; 0 Providers | 0; 0 Providers | 0; 0 Providers

BASELINE CHARACTERISTICS:
Population: There were 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads. The number of dyads is represented in the Overall Number of Baseline Participants above. Baseline Characteristics for both parents and children are represented below.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care | Total
Number analyzed (Participants) | 1422 | 1504 | 1154 | 4080
Age, Continuous [Mean (Standard Deviation); unit: Child Age (Months), mean (SD)] — Population: Only child age is represented.
  Child Age (Months), mean (SD)
    number analyzed (Participants) | 711 | 752 | 577 | 2040
    (all) | 35.8 (11.3) | 35.2 (11.2) | 35.4 (10.9) | 35.5 (11.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: There were 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads.
  Participants
    Sex of Child: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Sex of Child: Female | 333 | 388 | 269 | 990
    Sex of Child: Male | 378 | 364 | 308 | 1050
    Sex of Child: Unknown | 0 | 0 | 0 | 0
    Sex of Parent: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Sex of Parent: Female | 663 | 696 | 539 | 1898
    Sex of Parent: Male | 34 | 33 | 29 | 96
    Sex of Parent: Unknown | 14 | 23 | 9 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There were 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads.
  Participants
    Race of Child: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Race of Child: Black | 70 | 39 | 46 | 155
    Race of Child: White | 619 | 690 | 506 | 1815
    Race of Child: Other | 22 | 23 | 25 | 70
    Race of Child: Unknown | 0 | 0 | 0 | 0
    Race of Parent: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Race of Parent: Black | 61 | 20 | 31 | 112
    Race of Parent: White | 568 | 651 | 489 | 1708
    Race of Parent: Other | 65 | 51 | 42 | 158
    Race of Parent: Unknown | 17 | 30 | 15 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There were 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads.
  Participants
    Ethnicity of Child: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Ethnicity of Child: Hispanic | 97 | 78 | 63 | 238
    Ethnicity of Child: Non-Hispanic | 614 | 674 | 514 | 1802
    Ethnicity of Child: Unknown | 0 | 0 | 0 | 0
    Ethnicity of Parent: number analyzed (Participants) | 711 | 752 | 577 | 2040
    Ethnicity of Parent: Hispanic | 80 | 74 | 56 | 210
    Ethnicity of Parent: Non-Hispanic | 617 | 657 | 508 | 1782
    Ethnicity of Parent: Unknown | 14 | 21 | 13 | 48
Region of Enrollment [Number; unit: Parent/Child dyads] — Population: There were 2040 unique parents and 2040 unique children that combined to form 2040 parent/child dyads. Data in this section are represented at the dyad not individual level as all participants were required to live in the United States.
  Parent/Child dyads
    United States: number analyzed (Participants) | 711 | 752 | 577 | 2040
    United States | 711 | 752 | 577 | 2040
BMI z-score, mean (SD) [Mean (Standard Deviation); unit: Child BMI z-score] — A z-score of 0 represents the population mean. Higher z-scores represent worse outcomes. BMI z-score over >=1 indicates possible risk for overweight. Population: BMI z-score are only analyzed on children.
  Child BMI z-score
    number analyzed (Participants) | 711 | 752 | 577 | 2040
    (all) | 1.05 (1.30) | 0.92 (1.08) | 1.03 (1.31) | 1.0 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Difference in BMI Z-score, Based on WHO Growth Standards
Description: BMI values will be obtained from Geisinger clinical care visits, documented in the EHR and standardized or parent-reported. Values obtained at well child visits during the study period, ideally 12 months, 1 day apart will be utilized but values within a 9- to 18-month span of baseline to 1-year follow up may be used (e.g., 3 months pre-baseline WCV to 15 months post-baseline, baseline WCV to 18-months post-baseline, etc.) to assess the primary outcome. A z-score of 0 represents the population mean. Higher z-scores represent worse outcomes. BMI z-score over >=1 indicates possible risk for overweight.
Time Frame: 1-year
Measure: Mean (Standard Error); unit: BMI z-score
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 711 | 752 | 577
BMI z-score | 1.005 (0.068) | 0.881 (0.066) | 0.979 (0.073)

2. Secondary Outcome: United States Household Food Security Survey Module: Six-Item Short Form
Description: This questionnaire uses 6 items to provide a scale of food security of high food security to very low food security. Scoring: Responses of "often" or "sometimes" on questions Q1 and Q2, and "yes" on Q3, Q5, and Q6 are coded as affirmative (yes). Responses of "almost every month" and "some months but not every month" on Q4 are coded as affirmative (yes). The sum of affirmative responses to the six questions in the module is the household's raw score on the scale. Food security status is assigned as follows: Raw score 0-1-High or marginal food security (raw score 1 may be considered marginal food security, but a large proportion of households that would be measured as having marginal food security using the household or adult scale will have raw score zero on the six-item scale); Raw score 2-4-Low food security. Raw score 5-6-Very low food security. Percentage of participants with low or very low food security scores were reported.
Time Frame: 1-year
Population: Only participants completing the Food Security section of the1-year survey were included in the overall number of participants analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage Low or Very Low Food Security
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 566 | 594 | 462
Percentage Low or Very Low Food Security | 16.9 [13.8 to 20.5] | 18.4 [15.3 to 21.9] | 21.4 [17.6 to 25.8]

3. Secondary Outcome: Modified Version of Perceived Involvement in Care Scale
Description: The Modified Perceived Involvement in Care Scale (M-PICS) measures patients' perceptions of doctor-patient communication during the medical encounter. PICs includes 4 domains including 1-Health care provider information 2- Patient information 3- Patient decision making 4- Health care provider facilitation. The total score combines these 4 domains with a range from 20 poor-100 high reported at 12-month follow-up.
Time Frame: 1-year
Population: Only participants completing the M-PICS section of the1-year survey were included in the overall number of participants analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 581 | 605 | 475
score on a scale | 71.81 (0.72) | 71.99 (0.71) | 72.92 (0.77)

4. Secondary Outcome: Food Resource Management
Description: Nine items from the Cooking Matters Food Resource Management survey that assess 2 subscales (each scored on 1-5 item Likert scale)- Food Resource Management Practices (indicating the frequency with which respondents engaged in behaviors to maximize food resources) and Food Resource Management Confidence (extent to which participants showed self-confidence in shopping, preparing foods, and managing food resources on a budget). Higher scores indicate more frequent practices and greater confidence, respectively. There is not a summary score. The scoring for each subscale uses the average of items within that subscale.
Time Frame: 1-year
Population: Only participants completing the Food Resource Management section of the1-year survey were included in the overall number of participants analyzed.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 566 | 594 | 462
Units on a scale
  Food Resource Management Practices | 3.76 (0.04) | 3.74 (0.04) | 3.78 (0.04)
  Food Resource Management Confidence | 3.96 (0.05) | 3.93 (0.05) | 4.03 (0.05)

5. Other Pre Specified Outcome: Raw BMI
Description: Differences in raw BMI will be evaluated amongst study arms.
Time Frame: 1-year
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 711 | 752 | 577
kg/m2 | 16.952 (0.114) | 16.735 (0.112) | 16.967 (0.125)

6. Other Pre Specified Outcome: BMI Units Above the 50th Percentile (BMI50)
Description: Differences in BMI50 will be evaluated amongst study arms. We reported using mean number of BMI units from the population mean which is defined as the distance from the BMI for age and sex at the 50th %tile.
Time Frame: 1-year
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 711 | 752 | 577
kg/m^2 | 1.596 (0.114) | 1.373 (0.113) | 1.609 (0.126)

7. Other Pre Specified Outcome: Percentage of Children Overweight and Obese
Description: Evaluate the percentage of children overweight and obese at 1-year follow-up per CDC guidance and definitions.
Time Frame: 1-year
Measure: Number; unit: Percent of total population
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
Number analyzed (Participants) | 711 | 752 | 577
Percent of total population
  % Overweight | 40.52 | 41.25 | 41.54
  % Obese | 22.89 | 23.56 | 22.85

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no expected adverse and/or serious adverse events.
Arm/Group | Standard of Care | Patient Reported Outcome | Patient Reported Outcome + Food Care
All-Cause Mortality (participants affected / at risk) | 0/711 | 0/752 | 0/577
Serious Adverse Events (participants affected / at risk) | 0/711 | 0/752 | 0/577
Other Adverse Events (participants affected / at risk) | 0/711 | 0/752 | 0/577

LIMITATIONS AND CAVEATS:
Limitations: Internal threats to validity may have influenced results including the Hawthorne effect and regression to the mean.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04406441/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04406441/ICF_001.pdf